CLINICAL TRIAL: NCT03560674
Title: Evaluation of Knowledge- Attitude- Practice (KAP) of Intern Dentists in Emergency Management of Traumatic Dental Injuries in Primary Anterior Teeth: A Cross-sectional Study
Brief Title: Evaluation of Intern Dentists in Emergency Management of Traumatic Dental Injuries in Primary Anterior Teeth
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Abd El-Naby Hussien, Principal Investigator, Cairo University
Other Study IDs: CEBD-CU-2018-4-10
Record Dates: First submitted 2018-05-30; First posted 2018-06-18 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Traumatic Injury
Keywords: Dental trauma; emergency management; traumatic injures.
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aim to evaluate knowledge, attitude, and practice of intern dentistry in emergency management of traumatic dental injures in primary anterior teeth in children aged from 3-5 years old. Questionnaire survey will be designed to evaluate Knowledge - Attitude - and practice of intern dentists who met the eligibility criteria

DETAILED DESCRIPTION:
Questionnaire survey will be designed to evaluate Knowledge - Attitude - and practice of intern dentists toward different forms of traumatic dental injuries in primary anterior teeth in children aged from 3 to 5 years old.

ELIGIBILITY:
Inclusion Criteria:

* Intern dentists attending their internship in Faculty of Dentistry- Cairo University, other private university (Modern Science and Arts University- MSA).
* The intern dentists who agree to participate.
* Intern dentists who did not attend Pediatric Dentistry round, Endodontic round, Emergency round and Surgery round at Cairo University.
* Intern dentists irrespective of age and sex.

Ages: 22 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Dentists attending their internship in Cairo University and another private university (Modern Science and Arts University- MSA).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-04-15 (Estimated); Study Completion 2019-05-15 (Estimated)

PRIMARY OUTCOMES:
Knowledge, attitude and practice (KAP) of intern dentists | 1 year
  measured by Knowledge, attitude and practice Questionnaire and the measuring unit is Binary (yes, no)
Knowledge, attitude and practice (KAP) of intern dentists | 1 year
  measured by Knowledge, attitude and practice Questionnaire and the measuring unit is Multiple choice questions

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Ahmed, Principal Investigator — Cairo University
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided